CLINICAL TRIAL: NCT04881084
Title: Learning to Care: Exploring Empathy and Compassion Using Digital Narratives
Brief Title: Exploring Empathy and Compassion Using Digital Narratives
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 254043
Record Dates: First submitted 2021-04-12; First posted 2021-05-11 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Mental Disorders, Severe; Mental Illness; Stigma, Social; Compassion; Empathy
Keywords: Digital Narratives; Digital Testimonials; Digital Stories; Social Marketing; Fundraising campaigns; Stigma; Mental Illness
MeSH Terms: conditions — Mental Disorders; Social Stigma | interventions — Social Marketing

STUDY DESIGN:
Intervention Model Description: Two-armed, parallel-design, individually randomized trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital storytelling group (Group 1) (Experimental): Participants will be randomly assigned to the digital storytelling group (n = 40 participants; 20 Anglophone and 20 Francophone; ages 18-35). Participants will be asked to watch twenty-six digital storytelling videos which will be assessed using a between-subjects design.
  Interventions: Other: Digital storytelling group
- Social marketing/fundraising group (Group 2) (Active Comparator): Participants will be randomly assigned to the social marketing/fundraising group (n = 40 participants; 20 Anglophone and 20 Francophone; ages 18-35). Participants will be asked to watch twenty-six social marketing/fundraising videos which will be assessed using a between-subjects design.
  Interventions: Other: Social marketing/fundraising group

INTERVENTIONS:
Other: Digital storytelling group — Participants (intervention- group 1) will watch digital stories, short videos describing the experience of recovering from mental illness created as part of this project. Participants in the control group (group 2) will watch social marketing and/or fundraising campaigns on similar topics and complete a few questionnaires. The following standardized scales will be used: The Level of Familiarity Scale (LOF) (which will be used only before exposure to movies); Toronto Empathy Questionnaire (16 items; internal consistency coefficient .79; test-retest reliability coefficient .73), Compassionate Love Scale (21 items; Cronbach's alpha: .95; item-to-total correlations ranging from .46 to .81), Dispositional Positive Emotions Scale (DPES) (5 items; Cronbach's alpha for the compassion subscale: .80; inter-scale correlations: .44), Self-Stigma of Mental Illness Scale-Short Form (SSMIS-SF) (20 items; Cronbach's alpha: 0.91); Difference and Disdain Scales for Public Stigma (DDSPS) (9 items).
  Arms: Digital storytelling group (Group 1)
Other: Social marketing/fundraising group — Participants will be randomly assigned to the social marketing/fundraising group (n = 40 participants; 20 Anglophone and 20 Francophone; ages 18-35). Participants will be asked to watch twenty-six social marketing/fundraising videos which will be assessed using a between-subjects design.
  Arms: Social marketing/fundraising group (Group 2)

SUMMARY:
Stories of suffering and struggle are shared continuously through digital formats such as internet videos, news stories, social marketing, and fundraising campaigns. Digital stories are often created and shared to generate awareness about a problem, impart knowledge on contemporary issues, or promote compassion. The practice of sharing critical life events and insights provided by these experiences are valuable for tellers and the listeners alike for catharsis, healing, reconciliation, and connectiveness. Portrayals of mental suffering are a matter of cultural and social interest as new media products become available to the public. Studies published since the 1990s overwhelmingly conclude that formal media depictions are biased, promoting the stereotype that people who suffer emotionally are mentally ill, dangerous, violent, or insane. Various agencies, organizations, and corporations are actively working to provide alternative stories/narratives to mainstream media by means of video testimonials in social marketing and fundraising campaigns and, ultimately, by taking advantage of the Internet. The impact of this work is under-researched. However, preliminary evaluations of social marketing campaigns report mixed results and raise questions about their effectiveness. As well, the first-person narrative prepared digitally and shared online is also providing alternative narratives to mainstream media stories. People are increasingly using digital videos to share their stories, viewing this as an opportunity to understand their emotions and thoughts, come to terms with disgrace around sensitive, personal issues and marginalization while providing hope and encouragement to others. This proposed study focuses on the process of creating digital narratives/stories, especially stories of mental and emotional suffering, and their impact in terms of inciting empathy, compassion, and good citizenship among viewers.

DETAILED DESCRIPTION:
Digital stories -- first person, self-made 2-3-minute videos -- aim to generate awareness about problems, impart knowledge, or promote compassion. Sharing critical life events and related insights are invaluable for tellers and listeners alike, supporting catharsis, healing, reconciliation, and connectiveness. Digital stories are created and shared among organizations or citizens ( "ordinary" people without a background in filmmaking) to promote awareness of particular problems. They impact peoples' knowledge of contemporary issues, shaping attitudes by stimulating empathy, compassion, and active citizenship.

The proposed study explores digital stories/narratives, particularly those focused on mental health recovery, and how stories elicit empathy and compassion by addressing three main questions: (1) How is mental and emotional suffering depicted in video testimonies presented by social marketing/fundraising campaigns, versus the stories of ordinary people told through digital videos? (2) What impact does digital storytelling have for the creators, as ordinary people willing to revisit difficult life moments and transform them into digital videos? (3) What is the impact of video depictions on viewers in terms of empathy and compassion?

This mixed-method study has 3 phases: In Phase 1 (Preparation), a search will be conducted to identify activities related to Canadian social marketing and fundraising campaigns. Digital storytelling workshops will be held simultaneously, and in-depth interviews conducted before and after each workshop. Social service and community organizations located in Montreal, Canada, will be contacted to promote the digital storytelling workshops, to be implemented in the community and on university campuses. In Phase 2, a pilot randomized controlled trial (RCT) will be undertaken and more in-depth interviews conducted. Phase 3 will consist of knowledge dissemination activities.

The knowledge acquired through this study on individual and societal responses to stories of human suffering will have a practical impact on future social marketing campaigns promoted by government agencies, fundraising campaigns launched by nonprofit and for-profit organizations, and the public. Results will consolidate previous knowledge while providing new insights into what prompts citizens to help others.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years of age
* Not currently admitted to a hospital

Exclusion Criteria:

* Not in age range (18-35 years of age)
* Currently admitted to a hospital
* Attended the digital storytelling workshop and made a digital story used in the RCT

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Empathy | Baseline, immediately after the intervention
  Change in empathy using the Toronto Empathy Questionnaire. The minimum scoring value is 0 and the maximum scoring value is 64. A higher score means a better outcome.
Compassion | Baseline, immediately after the intervention
  Change in compassion using the Compassionate Love Scale. The minimum scoring value is 1 and the maximum scoring value is 7, which comes from the average of all item scores. A higher score means a better outcome.

SECONDARY OUTCOMES:
Positive emotions | Baseline, immediately after the intervention
  Change in positive emotions using the Dispositional Positive Emotions Scale. The minimum scoring value is 5 and the maximum scoring value is 35. A higher score means a better outcome.
Mental health self-stigma | Baseline, immediately after the intervention
  Change in mental health stigma using the Self-Stigma of Mental Illness Scale-Short Form. The minimum scoring value is 20 and the maximum scoring value is 180. A higher score means a worse outcome.
Mental health public stigma | Baseline, immediately after the intervention
  Change in mental health stigma using the Difference and Disdain Scales for Public Stigma. The minimum scoring value is 9 and the maximum scoring value is 81. A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferrari M, Fazeli S, Mitchell C, Shah J, Iyer SN. Exploring Empathy and Compassion Using Digital Narratives (the Learning to Care Project): Protocol for a Multiphase Mixed Methods Study. JMIR Res Protoc. 2022 Jan 13;11(1):e33525. doi: 10.2196/33525. PMID 35023844